CLINICAL TRIAL: NCT07295184
Title: Effect of Rebound Pain on Postoperative Intensive Care Delirium in Patients Undergoing Hip Surgery With Peripheral Nerve Block: A Prospective Observational Study
Brief Title: Effect of Rebound Pain on Postoperative Intensive Care Delirium in Patients Undergoing Hip Surgery With Peripheral Nerve Block
Status: Not yet recruiting | Type: Observational
Sponsor: Konya City Hospital (Other)
Responsible Party: Principal Investigator, HASAN ŞENAY, Specialist, Department of Intensive Care Unit, Konya City Hospital, M.D, Konya City Hospital
Other Study IDs: Rebound pain
Record Dates: First submitted 2025-12-08; First posted 2025-12-19 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Rebound Pain Impact After Hip Surgery With Nerve Block

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Peripheral nerve block applied — Pericapsular Nerve Group block and the supra-inguinal fascia iliaca block applied
Other: Only multimodal analgesia applied — Postoperative analgesia (paracetamol 1000 mg intravenously every 8 hours and celecoxib 200 mg orally every 12 hours)

SUMMARY:
Postoperative delirium is a significant and commonly encountered complication in patients undergoing hip surgery, particularly among the elderly. Postoperative delirium is associated with serious consequences, including prolonged intensive care unit stay, increased complication rates, higher mortality risk, and rising healthcare costs.

The incidence of Postoperative delirium after hip fracture surgery has been reported to range between 13% and 55.9%, indicating a substantial clinical burden.

Effective postoperative pain control is critical not only for maintaining quality of life but also for preserving cognitive well-being. In this context, peripheral nerve blocks are frequently used for pain management following hip surgery.

DETAILED DESCRIPTION:
Postoperative delirium is a significant and commonly encountered complication in patients undergoing hip surgery, particularly among the elderly. Postoperative delirium is associated with serious consequences, including prolonged intensive care unit stay, increased complication rates, higher mortality risk, and rising healthcare costs.

The incidence of Postoperative delirium after hip fracture surgery has been reported to range between 13% and 55.9%, indicating a substantial clinical burden.

Effective postoperative pain control is critical not only for maintaining quality of life but also for preserving cognitive well-being. In this context, peripheral nerve blocks are frequently used for pain management following hip surgery.

In recent years, the Pericapsular Nerve Group block and the supra-inguinal fascia iliaca block have gained attention as regional anesthesia techniques that provide effective analgesia by targeting the nerve branches innervating the anterior capsule of the hip joint.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-80
* ASA I-III risk groups
* Undergoing elective hip surgery

Exclusion Criteria:

* Preoperative history of delirium, dementia, or major neurological disease
* Present cognitive impairment or severe hearing or visual impairment that could affect pain assessment
* Development of mechanical ventilation requirement in the intensive care unit; Need for bilateral hip surgery
* Failure to provide meaningful analgesia after block application due to surgical pain outside the scope of the block
* Patient's inability to complete the pain diary during postoperative follow-up;
* Urgent hip surgery
* Voluntary failure to give consent or request to withdraw from the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We conducted a pilot study on 20 patients using the 'goodness-of-fit tests: contingency tables' test with G Power software. In our study, the incidence of rebound pain was 40%, and postoperative delirium developed in 50% of patients with rebound pain, compared to 8.3% in patients without rebound pain.
  Based on these data, an effect size of 0.356 was found, and an analysis was conducted using α=0.05, 90% power.
  The sample size was calculated as 83 patients. Considering the dropout rate, a total of 90 patients (36 patients with rebound pain and 54 patients without rebound pain) were calculated to be included in the study.
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2025-12-25 (Estimated); Primary Completion 2026-12-25 (Estimated); Study Completion 2026-12-25 (Estimated)

PRIMARY OUTCOMES:
Incidence of delirium | 72 hours
  The incidence of delirium will be evaluated in the first 72 hours postoperatively in the intensive care unit.